CLINICAL TRIAL: NCT03511092
Title: The Effects of β-hydroxy-β-methylbutyrate and Leucic Acid in Performance, Body Composition and Biochemical Markers
Brief Title: The Effects of Leucine Metabolites in Performance, Body Composition and Biochemical Markers of Muscle Damage
Acronym: LMET2IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Cristina Monteiro, Assistant Professor, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LabFisiolBioqMLeu
Record Dates: First submitted 2018-04-02; First posted 2018-04-27 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Resistance Training
Keywords: Leucine metabolites; Resistance training; Hypertrophy; Strength; Supplement
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HMB-FA (Experimental)
  Interventions: Dietary Supplement: HMB-FA
- HMB-Ca (Experimental)
  Interventions: Dietary Supplement: HMB-Ca
- alfa-HICA (Experimental)
  Interventions: Dietary Supplement: alfa-HICA
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Dietary Supplement: HMB-FA — One gram of HMB-FA was ingested before exercise, and two grams were ingested at subsequent meals (1 g per meal). At rest days supplement was administered 1 g per meal. The total duration of the intervention was 8 weeks.
  Arms: HMB-FA
Dietary Supplement: HMB-Ca — One gram of HMB-Ca was ingested before exercise, and two grams were ingested at subsequent meals (1 g per meal). At rest days supplement was administered 1 g per meal. The total duration of the intervention was 8 weeks.
  Arms: HMB-Ca
Dietary Supplement: alfa-HICA — Five hundred miligram of alfa-HICA was ingested before exercise, and one gram was ingested at subsequent meals (500 mg per meal). At rest days supplement was administered 500 mg per meal. The total duration of the intervention was 8 weeks.
  Arms: alfa-HICA
Other: Placebo comparator — One gram of magnesium stearate was ingested before exercise, and two grams were ingested at subsequent meals (1 g per meal). At rest days placebo was administered 1 g per meal. The total duration of the intervention was 8 weeks.
  Arms: Placebo

SUMMARY:
This study aimed to conduct a double-blind randomized pragmatic trial to evaluate the effects of off-the-shelf leucine metabolite supplements HMB-FA, HMB-Ca, alfa-HICA, on resistance training-induced changes in body composition, performance and biochemical markers of muscle damage. The investigators' working hypothesis is that so long as subjects adhered to a diet containing adequate energy and dietary protein, there would be no differences between those receiving the leucine metabolites - HMB-FA, HMB-Ca and alfa-HICA - when compared to a placebo consuming group.

DETAILED DESCRIPTION:
This was a randomized, double blind, placebo-controlled study with additional control of diet. The investigators compared the effect of 8 weeks of supplementation with HMB-FA, HMB-Ca, or alfa-HICA on performance, body composition, and biochemical markers of muscle damage. The study involved fifty-three participants engaged in resistance training for at least one year (≥3 training sessions per week).

Performance measures - To evaluate aerobic performance an incremental test to volitional exhaustion was performed. Peak power and strength was assessed by maximum strength and the participants also performed a Wingate and vertical jump tests. Perceived performance and recovery was measured by the perceived recovery status scores in training days. This tool allowed to evaluate both fatigue, general muscle soreness, sleep quality, stress levels and mood throughout the study. Performance tests were performed at baseline, prior to the beginning of the study, and at the end of weeks 4 and 8, in a fed state (a meal replacement bar was provided to participants before the tests).

Body composition measures - To evaluate body composition a dual-energy X-ray absorptiometry (DXA) scan was performed; Muscle thickness was measured by ultrasonography; Total body water and both the extracellular water and intracellular water were assessed by bioelectrical impedance spectroscopy (BIS). These tests were performed at baseline and at the end of weeks 4 and 8, with participants reporting to the lab in a fasted state, refraining from exercise, alcohol or stimulant beverages for at least 8 h.

Biochemical markers of muscle damage - To assess biochemical markers (total testosterone and cortisol, creatine kinase, insulin-like growth factor 1, growth hormone), blood was collected at baseline and at the end of weeks 4 and 8, in a fasted state with participants also refraining from exercise, alcohol or stimulant beverages for at least 12 h.

Training protocol - The training program was designed according to the guidelines for hypertrophy type of resistance training for intermediate-trained individuals and consisted on 3 sessions per week during an 8-week period.

Statistics - sample size was calculated through an a priori power analysis (G*Power Version 3.1.9.2, Heinrich Heine Universitat Dusseldorf, Germany), based on FFM changes from previous studies and power of 0.80. Statistical analysis will be performed using IBM SPSS statistics version 22.0 (IBM, Chicago, Illinois, USA). Normality of the distribution of variables will be tested by Shapiro-Wilk test. Baseline characteristics between groups were analyzed by a 1-way analysis of variance (ANOVA) since normality was observed. Time and time x group interactions will be evaluated by repeated-measures ANOVA. The equality of the matrix of variance and sphericity will be explored with the Levene F test and Mauchly's test, respectively. Overall significance level for α was set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Resistance training subjects for more than one year

Exclusion Criteria:

* Individuals taking any type of drug, medicines or supplements that may enhance body composition or performance, 1 months prior to the research.
* Smokers
* Clinical diagnose of a disease that might compromise tolerance to the supplements or influence body composition and performance
* More than 25% body fat
* Individuals involved in similar research 3 months prior to the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Change of maximum strength | Baseline, week 4 and week 8
  kg
Change of peak power | Baseline, week 4 and week 8
  Watt
Change of jump height | Baseline, week 4 and week 8
  cm
Change of power | Baseline, week 4 and week 8
  Watt
Change of muscle thickness | Baseline, week 4 and week 8
  mm
Change of fat free mass | Baseline, week 4 and week 8
  kg
Change of fat mass | Baseline, week 4 and week 8
Change of body water | Baseline, week 4 and week 8
  kg

SECONDARY OUTCOMES:
Change of biochemical markers of muscle damage | Baseline, week 4 and week 8
  total testosterone and cortisol, creatine kinase, insulin-like growth factor 1, growth hormone
Oxygen uptake | Baseline and week 8
  mL.kg-1.min-1
Heart rate | Baseline and week 8
  beats.min-1

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No